CLINICAL TRIAL: NCT02255357
Title: Investigation of the Effect of Intranasal Oxytocin on Relapse Risk in Cocaine-dependent Patients
Brief Title: Investigation of Intranasal Oxytocin on Relapse Risk in Cocaine-dependent Patients.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Wilfrid Raby, Principal Investigator, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #6933; DA035461-01A1 (Other Grant/Funding Number: NIDA)
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Results first posted 2019-11-29 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Cocaine Dependence
Keywords: Oxytocin; Vasopressin; Cocaine
MeSH Terms: conditions — Cocaine-Related Disorders; Diabetes Insipidus | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Solution containing only the excipients of the original solution without Oxytocin.
  Interventions: Drug: Placebo
- Intranasal Syntocinon (Active Comparator): Intranasal Oxytocin 24 IU per day.
  Interventions: Drug: Intranasal Oxytocin

INTERVENTIONS:
Drug: Placebo — Solution containing only the excipients of the original solution without Oxytocin.
  Arms: Placebo
Drug: Intranasal Oxytocin — solution containing Oxytocin 6 IU/0.1cc or per puff is used in this arm
  Other Names: Syntocinon
  Arms: Intranasal Syntocinon

SUMMARY:
This proposal describes a combined laboratory and clinical trial preliminary investigation to advance medication development for cocaine dependence. The main objective is to test whether intranasal Oxytocin could reduce relapse risk by reducing stress sensitivity. To measure the stress sensitivity, this study will evaluate a new stress challenge: a) Intranasal desmopressin, a vasopressin analog, will be used an endocrine stressor; its effects will be evaluated by serial measurements of serum Adrenocorticotropin hormone (ACTH), and self reports; b) if pretreatment with intranasal oxytocin dampens the ACTH and subjective response to intranasal desmopressin. These measures will be tested during a 7-day inpatient abstinence induction hospitalization. For those patients with family and work obligations, an outpatient abstinence induction procedure is available. The response to the desmopressin challenge will be compared to a cohort of matched control subjects. After abstinence induction, cocaine dependent patients enter a 6-week, double blind, randomized, placebo-controlled trial of 24 IU of intranasal oxytocin vs. placebo, to monitor if this reduces the relapse risk.

DETAILED DESCRIPTION:
This study is based on the findings that chronic stress, caused in these patients by cocaine dependence, increases the sensitivity of the Hypothalamo-Pituitary-Adrenal (HPA) axis and CNS stress pathways to vasopressin. For their part, oxytocin systems, in chronic stress, acquire an increasing moderating effect on CNS stress system and the HPA axis. Cocaine dependence generates increased responsivity of stress system to oxytocin in the face of depleted oxytocin stores; thus creating an environment where exogenous oxytocin could exert a strong regulatory effect. Intranasal administration provides a convenient method to deliver these small peptides to the brain. Studying the feasibility of this approach, and its applicability to the treatment of cocaine-dependent patients, will be a goal of the study. The main outcome of this study will be the number of consecutive days of abstinence from cocaine after abstinence induction. A secondary outcome will be: Is the acute effect of intranasal oxytocin on desmopressin-induced ACTH secretion associated with the number of days of continued abstinence.

ELIGIBILITY:
Study Inclusion Criteria (cocaine-dependent participants):

* Age 18 to 60.
* Meet DSM-IV criteria for current cocaine dependence and is seeking treatment.
* Displays at least one cocaine-positive urine toxicology during screening.
* Use of cocaine at least 4 days in the past month, with at least weekly use, or reports episodic binges of large amounts of cocaine (at least $200) at least 2x/month.
* Able to give informed consent and comply with study procedures.
* Can pass the blindfolded scent test recognizing the scent of cinnamon or coffee.

Study Exclusion Criteria (cocaine-dependent participants):

* Meets DSM-IV criteria for bipolar disorder, schizophrenia or any psychotic disorder other than transient psychosis due to drug abuse. Severe depression is an exclusion criteria (Hamilton Depression Scale ≥ 15).
* History of allergy or adverse event related to Oxytocin or Desmopressin. Patient using Oxytocin or Vasopressin-based products cannot participate.
* Chronic organic mental disorder, insufficient proficiency in English, or any condition or status (illiteracy) that would render an individual incapable of giving informed consent.
* Significant current suicidal risk, suicide attempt within the past year.
* Unstable physical disorders, which might make participation hazardous.
* Coronary Vascular disease as indicated by history, or suspected by abnormal ECG.
* Currently meets DSM-IV criteria for another substance dependence or abuse disorder other than nicotine, or alcohol. If alcohol dependent, must not be in need of detoxification.
* Participants who cannot comply with study procedures during the inpatient or outpatient abstinence induction (phase 1) will not proceed to Phase 2.
* Pregnancy, positive urine pregnancy test, or breastfeeding. Women who wish to participate must agree to use a method of contraception during the study and sign a written commitment to that effect, and submit to a urine pregnancy test every two weeks of Phase 2.
* History of transphenoidal surgery or sinus surgery in the past month. Simple nasal congestion is not exclusionary.

Study Inclusion Criteria (healthy volunteers):

* Age 18 to 60.
* Able to give informed consent and comply with study procedures.
* Can pass the blindfolded scent test recognizing the scent of cinnamon or coffee.

Study Exclusion Criteria (healthy volunteers):

* DSM-IV Axis 1 psychiatric diagnosis. Severe Major Depression (Hamilton Depression Scale > 15) is an exclusion criteria.
* Unstable physical disorders, which might make participation hazardous.
* Diagnosis of Substance Abuse or Dependence disorder, with exception of nicotine dependence. Patients in remission may participate if its duration is greater than 2 years preceding participation.
* History of allergy or adverse event related to oxytocin or desmopressin. Patient using oxytocin or vasopressin-based products cannot participate.
* Chronic organic mental disorder, insufficient proficiency in English or illiteracy that would render an individual incapable of giving informed consent.
* History of transphenoidal surgery or sinus surgery in the past month. Simple nasal congestion is not exclusionary.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2015-03; Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilfrid N Raby, PhD, MD, Principal Investigator — Division of Substance Abuse, Department of Psychiatry - Columbia university
Locations (2):
- United States (2):
  - Substance Treatment and Research Service (STARS), Manhattan, New York
  - Divison on Substance Abuse - Albert Einstein College of Medicine, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Araya AV, Rojas P, Fritsch R, Rojas R, Herrera L, Rojas G, Gatica H, Silva H, Fiedler JL. Early response to venlafaxine antidepressant correlates with lower ACTH levels prior to pharmacological treatment. Endocrine. 2006 Dec;30(3):289-98. doi: 10.1007/s12020-006-0007-2. PMID 17526941
- [Background] Manning M, Stoev S, Chini B, Durroux T, Mouillac B, Guillon G. Peptide and non-peptide agonists and antagonists for the vasopressin and oxytocin V1a, V1b, V2 and OT receptors: research tools and potential therapeutic agents. Prog Brain Res. 2008;170:473-512. doi: 10.1016/S0079-6123(08)00437-8. PMID 18655903
- [Background] Rodrigues SM, Saslow LR, Garcia N, John OP, Keltner D. Oxytocin receptor genetic variation relates to empathy and stress reactivity in humans. Proc Natl Acad Sci U S A. 2009 Dec 15;106(50):21437-41. doi: 10.1073/pnas.0909579106. Epub 2009 Nov 23. PMID 19934046
- [Background] Suzuki Y, Yamamoto S, Umegaki H, Onishi J, Mogi N, Fujishiro H, Iguchi A. Smell identification test as an indicator for cognitive impairment in Alzheimer's disease. Int J Geriatr Psychiatry. 2004 Aug;19(8):727-33. doi: 10.1002/gps.1161. PMID 15290695
- [Background] Weiss RD, Griffin ML, Hufford C, Muenz LR, Najavits LM, Jansson SB, Kogan J, Thompson HJ. Early prediction of initiation of abstinence from cocaine. Use of a craving questionnaire. Am J Addict. 1997 Summer;6(3):224-31. PMID 9256988
- See also: Oxytocin description — http://www.pdr.net/drug-summary/pitocin?druglabelid=1666&mode=preview
- See also: Desmopressin Acetate description — http://www.pdr.net/drug-summary/ddavp-nasal-spray?druglabelid=1034&mode=preview

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For control participants, reasons for not being included in the final analysis included: 1) not completing the laboratory protocol (phase 1) the only portion of the study that they participated in. 2 did not complete, and 1 was excluded for medical complication during the laboratory challenge.
  For Cocaine use disorder patients, reasons for not included in the analysis or not counting as completers: 1) droping out after the initial inpatient laboratory phase;
Period: Overall Study
Arm/Group | Placebo | Intranasal Syntocinon
Started | 14 | 29
Completed | 4 | 5
Not Completed | 10 | 24
Not completed — Physician Decision | 10 | 24

BASELINE CHARACTERISTICS:
Population: Placebo patients receive IN placebo solution, 2 insufflations per nostril, those randomized to Intranasal Oxytocin receive daily insufflation of 24 IU, or 2 insuflations per nostril.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Intranasal Syntocinon | Total
Number analyzed (Participants) | 14 | 29 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 29 | 43
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 13
  Male | 11 | 19 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 27 | 40
  White | 0 | 0 | 0
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 29 | 43

OUTCOME MEASURES:

1. Primary Outcome: Weeks of Abstinence From Cocaine
Description: this is outcome for the phase 2, clinicial trial portion of this combined laboratory and clinical trial laboratory human study
  For the human laboratory study, Phase 1, the primary outcome is differences in ACTH levels following a) Intranasal Desmopressin, and, on a consecutive day, b) Intranasal Desmopressin preceded by a treatment with Intranasal Oxytocin (Syntocinon). this takes place on 2 consecutive days
Time Frame: Phase 1: 7 days; Phase 2: 6 weeks
Measure: Mean (95% Confidence Interval); unit: weeks
Groups:
- Placebo for Phase 2, Clinical Trial: Solution containing only the excipients of the original solution without Oxytocin.
  Placebo: Solution containing only the excipients of the original solution without Oxytocin.
- Intranasal Syntocinon for Clinical Trial Phase 2: Intranasal Oxytocin 24 IU per day.
  Intranasal Oxytocin: solution containing Oxytocin 6 IU/0.1cc or per puff is used in this arm
Arm/Group | Placebo for Phase 2, Clinical Trial | Intranasal Syntocinon for Clinical Trial Phase 2
Number analyzed (Participants) | 14 | 29
weeks | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0]

ADVERSE EVENTS:
Time Frame: 6 months during randomized trial or participants length of participation
Arm/Group | Placebo | Intranasal Syntocinon
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/15
Other Adverse Events (participants affected / at risk) | 6/11 | 5/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | Intranasal Syntocinon (N=15)
feeling woozy (General disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
headache (General disorders) | 3 (3) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
feeling energized (General disorders) | 0 (0) | 3 (3)
less irritable (General disorders) | 0 (0) | 1 (1)
calm (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2014-09-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT02255357/Prot_000.pdf
  • Statistical Analysis Plan (2013-03-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT02255357/SAP_001.pdf